CLINICAL TRIAL: NCT01359072
Title: Enhancing Coping Skills in Patients With Cancer - a Randomized Controlled Study
Brief Title: Enhancing Coping Skills in Patients With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is currently terminated due to low recruitment rate.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Louise Granofsky-Psychosocial Oncology Program, Segal Cancer Centre, Montreal (Unknown)
Responsible Party: Principal Investigator, Dr. Annett Korner, PhD, Associate Member, Psychosocial Oncology Program, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-327-PSY
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Cancer
Keywords: coping; psychological distress; self-administered intervention
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention Treatment (Experimental)
  Interventions: Other: Self administered coping intervention
- Wait list (Experimental)
  Interventions: Other: Self administered coping intervention

INTERVENTIONS:
Other: Self administered coping intervention — The self administered coping intervention (i.e. NUCARE workbook) aims to teach individuals how to cope with their cancer. The intervention embraces two major areas: (i) the enhancement of a sense of personal control; and (ii) the learning of emotional and instrumental coping responses. The approach emphasizes training in problem-solving, relaxation techniques, cognitive coping skills, goal setting, communication, social support and lifestyle factors. The didactic material of the Nucare program is comprised of a workbook containing 12 chapters addressing the above mentioned aspects.

SUMMARY:
* Approximately 30% of all patients with cancer report levels of psychological distress indicative of the need for psychological intervention.
* Research suggests that learning more adaptive coping strategies improves psychological adjustment to cancer.
* It is imperative to develop cost-efficient, feasible psychosocial interventions.
* The aim is to test the efficacy of the self administered format of a psycho-educational intervention (NUCARE) in reducing distress and enhancing adaptive coping strategies for cancer patients.

It is hypothesized that:

* patients would show significant reductions in distress (i.e., depression and anxiety) over the 6-week treatment period, and that treatment would produce superior results compared to wait-list; patients would maintain or even increase their improvement up to 3 months following treatment.
* the treatment would enhance more adaptive coping strategies.
* greater self-reported adherence to the treatment/homework would be associated with symptom improvement, more autonomous self-regulation and higher perceived competence for adhering to the coping intervention program.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age,
* able to read English,
* a cancer patient presenting at the McGill University Health Centre (MUHC) interested in participating,
* willing to receive minimal therapist contact (by telephone) and self administered therapy,
* able to give their own consent.

Exclusion Criteria:

* currently receiving psychological/psychiatric treatment/counselling,
* indicate at the time of recruitment that they intend to seek psychological treatment elsewhere during the study period,
* a history of psychosis or bipolar disorder,
* substance abuse/dependence in last 6 months,
* taking psychotropic medication with altering dosages in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in The Health Education Impact Questionnaire from pre to post intervention, at 6 weeks post intervention, and 3 months post intervention | pre-intervention (week 0), post intervention (week 6), 6 weeks post intervention, 3 months post intervention

SECONDARY OUTCOMES:
Change in coping strategies & distress from pre to post intervention, at 6 weeks post intervention, and 3 months post intervention | pre-intervention (week 0), post intervention (week 6), 6 week post intervention, 3 month post intervention
  Measured with The Ways of Coping Questionnaire - Cancer Version scale and the Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Annett Koerner, PhD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre - Melanoma Clinic & Cedars CanSupport, Montreal, Quebec, Canada